CLINICAL TRIAL: NCT06255821
Title: The Effect of Time on Generalization of Exposure-based Benefit in Spider Fear
Brief Title: The Effect of Time on Generalization of Exposure-based Benefit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Iris Kodzaga, Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ruhr-University Bochum
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2024-07

CONDITIONS: One Week Follow-up Assessment; Six Weeks Follow-up Assessment; Three Months Follow-up Assessment
Keywords: Exposure Therapy; Generalization of Exposure Effects; Fear of Spiders; Anxiety Disorders; Extinction; Specific phobia
MeSH Terms: conditions — Arachnophobia; Anxiety Disorders; Phobia, Specific

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One week follow-up assessment (Experimental): Participants will receive a pre-assessment and an exposure with a control spider (spider A). This control spider will be presented again at post-training assessments. Participants will then be assigned to the follow-up assessment one week after the exposure session, in which spider A and a novel spider (spider B) will be used to test for generalization of exposure effects.
  Interventions: Behavioral: Exposure
- Six weeks follow-up assessment (Experimental): Participants will receive a pre-assessment and an exposure with a control spider (spider A). This control spider will be presented again at post-training assessments. Participants will then be assigned to the follow-up assessment six weeks after the exposure session, in which spider A and a novel spider (spider B) will be used to test for generalization of exposure effects.
  Interventions: Behavioral: Exposure
- Three months follow-up assessment (Experimental): Participants will receive a pre-assessment and an exposure with a control spider (spider A). This control spider will be presented again at post-training assessments. Participants will then be assigned to the follow-up assessment three months after the exposure session, in which spider A and a novel spider (spider B) will be used to test for generalization of exposure effects.
  Interventions: Behavioral: Exposure

INTERVENTIONS:
Behavioral: Exposure — One-session of graded in-vivo exposure with a spider. Each task is first modeled by the experimenter. Prior to the exposure, participants receive psychoeducation on anxiety and phobias.

SUMMARY:
Participants will receive a pre-assessment and an exposure with a control spider. This control spider will be presented again at post-training assessments. Participants will then be assigned to one of the follow-up assessments: one week, six weeks or three months. The control spider (spider A) and a novel spider (spider B) will be used again at follow-up BATs to test for generalization of exposure effects.

DETAILED DESCRIPTION:
Several findings from basic research on extinction learning undermine the role of time effects in the contextualization and retrieval of extinguished memories (Archbold et al., 2013; Quirk, 2002; Wiltgen & Silva, 2007). The latter bears important implications for the evaluation of short- and long-term effects of exposure-based fear reduction and generalization. To date, no study exists examining the role of time on the fear responding to treated stimuli and/or untreated stimuli after successful exposure. It will be investigated whether the differential responding to treated and untreated stimuli after exposure is dependent on the passage of time.

Spider fearful participants will be subjected to a standardized one-session treatment with spiders serving as treatment stimuli. Fear reduction towards treatment stimuli will be assessed at post-treatment. Furthermore, generalization of exposure therapy towards untreated stimuli (i.e., a novel spider) will be assessed. The extent of generalization of exposure-based fear reduction to untreated stimuli will be compared between three groups that will differ with respect to the follow-up length. Here, participants undergoing exposure will be randomly assigned to one of the following follow-up measurements: one week follow-up, six weeks follow-up, and three months follow-up. The extent of exposure induced fear reduction and generalization will be assessed and compared between these groups.

ELIGIBILITY:
Inclusion Criteria:

* Presence of fear of spiders (Potential diagnosis of arachnophobia)

Exclusion Criteria:

* Reaching level 10 or higher in the initial (Pre-Exposure) Spider BAT
* Any acute or chronic mental and / or somatic disease
* Psychological, psychiatric, neurological or pharmacological treatment
* Drug or alcohol abuse
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Behavioral Approach Test (BAT) | Pre-assessment (immediately before exposure), post-assessment (one day after exposure), follow-up (one week, six weeks, or three months after exposure)
  Change in the Behavioral Approach Test (BAT) at post-assessment and follow-up with the control spider (spider A; treated stimulus) and a novel spider (spider B; untreated fear stimulus). During the Behavioral Approach Test (BAT) the closest distance to a spider is measured.
Subjective fear | Pre-assessment (immediately before exposure), post-assessment (one day after exposure), follow-up (one week, six weeks, or three months after exposure)
  Change in subjective fear at post-assessment and follow-up with the control spider (spider A; treated stimulus) and a novel spider (spider B; untreated fear stimulus) is measured during the Behavioral Approach Tests.
Subjective disgust | Pre-assessment (immediately before exposure), post-assessment (one day after exposure), follow-up (one week, six weeks, or three months after exposure)
  Change in subjective disgust at post-assessment and follow-up with the control spider (spider A; treated stimulus) and a novel spider (spider B; untreated fear stimulus) is measured during the Behavioral Approach Tests.
Heart rate | Pre-assessment (immediately before exposure), post-assessment (one day after exposure), follow-up (one week, six weeks, or three months after exposure)
  Change in heart rate at post-assessment and follow-up with the control spider (spider A; treated stimulus) and a novel spider (spider B; untreated fear stimulus) is measured during the Behavioral Approach Tests.

SECONDARY OUTCOMES:
Score on General Self-efficacy (GSE) Scale | Pre-assessment (immediately before exposure), post-assessment (one day after exposure), follow-up (one week, six weeks, or three months after exposure)
  Change in self-efficacy is measured by the GSE Scale. The GSE Scale contains ten items and measures how confident the person feels to overcome difficult situations based on their self-assessed competence. The total score is determined by summing up all item scores, which results in a score between 10 and 40, where the higher scores represent higher GSE.
Self-efficacy Questionnaire for Phobic Situations (SEQ-SP) | Pre-assessment (immediately before exposure), post-assessment (one day after exposure), follow-up (one week, six weeks, or three months after exposure)
  The questionnaire consists of 13 items. The items describe specific phobic situations (in relation to animals) for which the participants has to assess their self-efficacy expectations based on a five-point scale (1 = really sure I couldn't, 5 = really sure I could).
Fear of Spiders Questionnaire (FSQ) | Pre-assessment (immediately before exposure), post-assessment (one day after exposure), follow-up (one week, six weeks, or three months after exposure)
  Change in the Spider-fear related questionnaires. The Fear of Spiders Questionnaire (FSQ) will be applied. Scores on this scale range from 0 to 108, with higher scores indicating greater fear of spiders.
Spider Fear Questionnaire (SPQ) | Pre-assessment (immediately before exposure), post-assessment (one day after exposure), follow-up (one week, six weeks, or three months after exposure)
  The Spider Fear Questionnaire (SPQ) will be applied. Scores on this scale range from 0 to 31, with higher scores indicating greater fear of spiders.
Spider Beliefs Questionnaire (SBQ) | Pre-assessment (immediately before exposure), post-assessment (one day after exposure), follow-up (one week, six weeks, or three months after exposure)
  The Spider Beliefs Questionnaire (SBQ) will be applied. Scores on this scale range from 0 to 100, with higher scores indicating greater fear of spiders.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Behavioral and Clinical Neuroscience, Bochum, Germany

IPD SHARING:
Plan to Share IPD: No